CLINICAL TRIAL: NCT03674151
Title: Randomized-controlled Trial of Wound Healing, Pain, Microbiology, Handling and Thrift of Different Wound Dressings in Patients With Split-skin Grafted Third Degree Burns
Brief Title: Trial of Different Wound Dressings in Split-skin Grafted Third Degree Burns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Luebeck (Other)
Responsible Party: Principal Investigator, Tobias Kisch, Principal Investigator, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-145-2
Record Dates: First submitted 2017-01-28; First posted 2018-09-17 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Split-skin Grafted Third-degree Burn Wound
Keywords: split-skin; burn wound; wound dressing; comparison; silver; honey; PVP-Iod; hydrogel
MeSH Terms: conditions — Burns | interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Device: Silver Nylon dressing (Active Comparator): 1/4 of a split-skin grafted third-degree burn wound in a Group (n=20): Consent-capable male and female patients ≥18 years of age who have a split-skin grafted third-degree burn on ≥3% and ≤30% of the surface of the body.
  Interventions: Device: Silver Nylon dressing
- Device: Manuka-Honey (Active Comparator): 1/4 of a split-skin grafted third-degree burn wound in a Group (n=20): Consent-capable male and female patients ≥18 years of age who have a split-skin grafted third-degree burn on ≥3% and ≤30% of the surface of the body.
  Interventions: Device: Manuka-Honey
- Device: Povidone-Iod (PVP-Iod) (Active Comparator): 1/4 of a split-skin grafted third-degree burn wound in a Group (n=20): Consent-capable male and female patients ≥18 years of age who have a split-skin grafted third-degree burn on ≥3% and ≤30% of the surface of the body.
  Interventions: Device: Povidone-Iod (PVP-Iod)
- Device: Hydrogel (Active Comparator): 1/4 of a split-skin grafted third-degree burn wound in a Group (n=20): Consent-capable male and female patients ≥18 years of age who have a split-skin grafted third-degree burn on ≥3% and ≤30% of the surface of the body.
  Interventions: Device: Hydrogel

INTERVENTIONS:
Device: Silver Nylon dressing — Non-staining Silver Nylon dressing with a permanently plated metallic surface on split-skin grafted third-degree burn wound
  Arms: Device: Silver Nylon dressing
Device: Manuka-Honey — Manuka-Honey dressing on split-skin grafted third-degree burn wound
  Arms: Device: Manuka-Honey
Device: Povidone-Iod (PVP-Iod) — Povidone-Iod (PVP-Iod) dressing on split-skin grafted third-degree burn wound
  Arms: Device: Povidone-Iod (PVP-Iod)
Device: Hydrogel — Hydrogel dressing on split-skin grafted third-degree burn wound
  Arms: Device: Hydrogel

SUMMARY:
In plastic and reconstructive surgery, treatment strategies of second-degree burn wounds and split-skin grafted third-degree burn wounds aim at reducing infection and improving reepithelialization. Although previous studies indicate that burn patients benefit from newer wound dressings, only a few studies comparing different wound dressings can be found. Therefore, the aim of this study is to evaluate time to reepithelialization, pain, microbiology, handling and costs of different wound dressings in patients with split-skin grafted third-degree burn wounds.

DETAILED DESCRIPTION:
In the treatment of burn wounds polyhexanide and betaisodona (PVP-Iod) are regularly used today. They act as antiseptics, but both have drawbacks. Polyhexanide evaporates fast and therefore cools patients when applied to a large wound area. Moreover, it is known to reveal a gap for pseudomonas. On the other hand, the half-life of Betaisodona (PVP-Iod) ranges between several minutes and 12 hours. Further, its application causes intense pain, and it is cytotoxic. Other wound dressings involving silver are frequently used, too. However, they color the wounds, which might therefore not be properly assessed. Silver is also thought to be cytotoxic.

New innovations are available today. In wound dressings with bound Silver ions wounds are not colored. Hydrolytic membranes keep the level of acidity low (acidic) and have therefore antiseptic effects that last until epithelialization of a second-degree burn wounds is completed. Medical honey is used in the treatment of chronic wounds and especially in pediatric surgery and oncology. Manuka honey from New Zealand is sterilized before application and is known to be less painful for the patient. Due to its acidic effect, it reduces germ numbers in the wounds. Honey can be left on the wound for more than one day, as well as hydrogel, that is also used for contaminated wounds.

These new wound dressings are just used in a couple of Burn Units for the treatment of second-degree burns or split-skin grafted burns. However, the treatment of large burn wounds with older dressing regimes (e.g. PVP-Iod) cause intensive pain in every dressing change.

Only a few studies pointing at new dressings in burn wounds can be found in the literature. None of them reveals a high quality randomized trial.

The objective of this clinical investigation is a direct comparison of established and newer wound dressings with respect to epithelialization time, pain and the number of pathogenic microbe species. Besides, handling and cost are analyzed.

This is a prospective, randomised, factorial, open clinical study. Endpoint assessment, primarily the time to epithelialization, for direct comparison of the dressings is performed in a blinded way. The aim of this study is to identify the advantages of each dressing.

Every wound dressing will be used in every patient. The order from proximal to distal is varied so that every dressing is at every position in a balanced number of cases and has the same neighbor dressing in a balanced number of cases (Williams-Design). The order is assigned by randomisation. All comparisons of two wound dressing can be made using the same number of paired observations.

Assessors of epithelialization time and germ burden are blinded to the wound dressing used.

ELIGIBILITY:
Inclusion Criteria:

* Consent-capable male and female patients
* ≥18 years of age
* ≥3% and ≤30% total body surface area (TBSA) split-skin grafted third-degree burn
* appropriate form of wound (not: too small) and localization (not: face, inplane surface)
* ability to asses pain

Exclusion Criteria:

* Immunosuppressive Therapy
* Clinical wound infection
* Allergy against porcine material, bee poison or honey, etherial oil, propyleneglycol, silver, nylon
* Relationship to someone who is involved in the study design or assessment
* Participation in other clinical trials
* Citizen of countries outside Europe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Epithelialization | through study completion, an average of 1 year
  Percent of epithelialized area

SECONDARY OUTCOMES:
Pain (on a visual analogue scale 0-10) | through study completion, an average of 1 year
  Assessed by VAS (visual analogue scale). 0 means no pain, 10 means maximum pain.
Microbiologic Smear | through study completion, an average of 1 year
  Assessed by gram staining and count
Subjective Handling | through study completion, an average of 1 year
  Assessed by rating scale (0-5)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kisch, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No